CLINICAL TRIAL: NCT03643250
Title: Lunch Feeding Study for Preschool Children
Brief Title: Effects of Varying Portion Size and Palatability on Food Intake of Preschool Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We observed reduced intake by the fifth week, so we are shortening the study and simplifying it by using a complete factorial design with four conditions.
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ChildFood401; R01DK082580 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Smaller Portion Size and Standard Appeal (non-divided plate) (Experimental): Food with Smaller Portion Size and Standard Appeal on a non-divided plate
  Interventions: Other: Smaller Portion Size and Standard Appeal (non-divided plate)
- Smaller Portion Size and Enhanced Appeal (divided plate) (Experimental): Food with Smaller Portion Size and Enhanced Appeal on a divided plate
  Interventions: Other: Smaller Portion Size and Enhanced Appeal (divided plate)
- Larger Portion Size and Standard Appeal (non-divided plate) (Experimental): Food with Larger Portion Size and Standard Appeal on a non-divided plate
  Interventions: Other: Larger Portion Size and Standard Appeal (non-divided plate)
- Larger Portion Size and Enhanced Appeal (divided plate) (Experimental): Food with Larger Portion Size and Enhanced Appeal on a divided plate
  Interventions: Other: Larger Portion Size and Enhanced Appeal (divided plate)
- Smaller Portion Size and Standard Appeal (divided plate) (Experimental): Food with Smaller Portion Size and Standard Appeal on a divided plate
  Interventions: Other: Smaller Portion Size and Standard Appeal (divided plate)

INTERVENTIONS:
Other: Smaller Portion Size and Standard Appeal (non-divided plate) — Food with Smaller Portion Size and Standard Appeal on a non-divided plate
  Arms: Smaller Portion Size and Standard Appeal (non-divided plate)
Other: Smaller Portion Size and Enhanced Appeal (divided plate) — Food with Smaller Portion Size and Enhanced Appeal on a divided plate
  Arms: Smaller Portion Size and Enhanced Appeal (divided plate)
Other: Larger Portion Size and Standard Appeal (non-divided plate) — Food with Larger Portion Size and Standard Appeal on a non-divided plate
  Arms: Larger Portion Size and Standard Appeal (non-divided plate)
Other: Larger Portion Size and Enhanced Appeal (divided plate) — Food with Larger Portion Size and Enhanced Appeal on a divided plate
  Arms: Larger Portion Size and Enhanced Appeal (divided plate)
Other: Smaller Portion Size and Standard Appeal (divided plate) — Food with Smaller Portion Size and Standard Appeal on a divided plate
  Arms: Smaller Portion Size and Standard Appeal (divided plate)

SUMMARY:
The aim of the study is to determine the effect of varying both the portion size and the appeal (palatability and presentation) of foods served to preschool children at a meal on the outcomes of food and energy intake at the meal.

ELIGIBILITY:
Inclusion Criteria:

* Children who are enrolled in a scheduled classroom of the designated childcare centers

Exclusion Criteria:

* Children who are allergic to any of the foods served
* Children whose diets exclude any of the foods served
* Children who will not be present at the childcare center for all of the scheduled study days

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Difference between interventions in meal energy intake | Study weeks 1, 2, 3, 4, and 5
  Energy consumed at the meal (kcal)

SECONDARY OUTCOMES:
Difference between interventions in food intake | Study weeks 1, 2, 3, 4, and 5
  Weight of food consumed at the meal (g)
Difference between interventions in meal energy density | Study weeks 1, 2, 3, 4, and 5
  Energy density of the food consumed at the meal (kcal/g)

OTHER OUTCOMES:
Liking of food served at the meal | Study week 6
  The Yummy-Yucky Cartoon Faces Scale (1=Yucky, 2=Just Okay, and 3=Yummy)
Preference of plate and vegetables served at the meal | Study week 6
  Preferred version of plate (1=non-divided plate, 2=divided plate), broccoli (1=standard appeal, 2=enhanced appeal), and corn (1=standard appeal, 2=enhanced appeal) of the two versions presented

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for the Study of Human Ingestive Behavior, The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No